CLINICAL TRIAL: NCT02226055
Title: An Investigation Into the Cardiovascular Risk and Aetiology of CKDu in Sri Lanka
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Rajarata University, Sri Lanka (Other)
Responsible Party: Sponsor
Other Study IDs: UoECKDu1
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: CKDu; Arterial Stiffness; Proteinuria; Serum Creatinine; Urinary Biomarkers; DNA Adducts
Keywords: Chronic kidney disease of unknown origin; Chronic kidney disease of unknown aetiology; Sri Lanka; CKDu; Arterial stiffness; Cardiovascular risk; North Central Province
MeSH Terms: conditions — Proteinuria | interventions — Pulse Wave Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urine samples: up to 30ml Blood samples: up to 40ml - 2 x EDTA blood bottles + 2 x serum gel Z bottles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Arterial stiffness: CKDu patients: Cohort of 50 patients with CKD of unknown aetiology Inclusion and exclusion criteria below Measure of arterial stiffness using pulse wave velocity technology Assessment of BMI, central and brachial blood pressure, arterial stiffness and 'arterial age' will be made and fed back to the patient. this information will be given in a 'results sheet' that the participant will be encouraged to give to their Gp for further treatments required.
  Interventions: Device: Arterial Stiffness Assessment
- Arterial stiffness: CKD known cause: Cohort of 50 patients with CKD of known cause Inclusion and exclusion criteria below Measure of arterial stiffness using pulse wave velocity technology Assessment of BMI, central and brachial blood pressure, arterial stiffness and 'arterial age' will be made and fed back to the patient. this information will be given in a 'results sheet' that the participant will be encouraged to give to their Gp for further treatments required.
  Interventions: Device: Arterial Stiffness Assessment
- Arterial Stiffness: Healthy Sri Lankan volunteers: Cohort of 50 participants who are healthy Sri Lankan volunteers Inclusion and exclusion criteria below Measure of arterial stiffness using pulse wave velocity technology Assessment of BMI, central and brachial blood pressure, arterial stiffness and 'arterial age' will be made and fed back to the patient. this information will be given in a 'results sheet' that the participant will be encouraged to give to their Gp for further treatments required.
  Interventions: Device: Arterial Stiffness Assessment
- 2nd aim: 250 CKDu patients for investigation of aetiology: To recruit a cohort of up to 250 CKDu patients from specific CKDu clinics in Anuradhapura and Padavi-Sri Pura for detailed history, basic anthropometric tests, and further analysis of serum, and urine. Analysis for biomarkers of kidney damage, proteomics, exosomes, and DNA adducts will be used to seek information that may complement already collected data and help refine aetiological hypotheses.
  Inclusion and Exclusion criteria as per CKDu cases in cohort 1

INTERVENTIONS:
Device: Arterial Stiffness Assessment — The following will be measured: brachial systolic and diastolic bp, heart rate, mean arterial bp, pulse pressure, brachial augmentation index (difference between the amplitudes of the late (backward) systolic wave (P2) and the early (forward) systolic wave (P1) over the pulse pressure x 100), central augmentation, ejection duration of the left ventricle, return time (time of the pulse wave travelling from aortic root to the bifurcation and back), aortic pulse wave velocity ( velocity of the pulse wave in the aorta), central systolic bp, central pulse pressure and diastolic reflection area (provides information about the quality of diastolic filling in the coronary arteries).
  We will perform an arterial age assessment. Patients are given a feedback form with their results to give to their general. Those with increased arterial stiffness will be tested for serum calcium and phosphate levels, and audited to ensure that a statin is commenced if not contraindicated.
  Other Names: TensioMed® Arteriograph™; Pulse wave velocity; Arterial Stiffness Monitor
  Groups: Arterial Stiffness: Healthy Sri Lankan volunteers; Arterial stiffness: CKD known cause; Arterial stiffness: CKDu patients

SUMMARY:
1. We hypothesise that CKDu patients will have increased arterial stiffness and thus increased all-cause and cardiovascular mortality. The first objective of this study is to recruit a cohort of ~ 50 CKDu patients who attend the CKDu clinic in Anuradhapura, and measure their arterial stiffness using the TensioMed® Arteriograph™ (details below). We will recruit an age, sex and blood pressure matched control group of healthy Sri Lankans (consenting visitors with patients both to clinic and as inpatients), and if possible, a second control group, similarly age, sex and blood pressure matched, who have CKD of known causes and attend general renal clinic in Anuradhapura.
2. We hypothesise that detailed renal analysis will give insight into the aetiology of CKDu in the North Central Province of Sri Lanka. The second objective of the study is to recruit up to 250 CKDu patients and to characterize their disease profile using analysis serum and urine renal biomarkers, exosomes, proteomics and DNA adducts.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is one of the leading causes of hospital admission, clinic attendance and mortality in some provinces of Sri Lanka. In central and southern provinces increased incidence is attributed to type-2 diabetes and hypertension; however, this is not the case in North Central Province (NCP) where CKD of unknown aetiology (CKDu) is the commonest diagnosis. A recent World Health Organisation (WHO) investigation concluded that at least 8,000 people have CKDu2.

First recognized in the early nineties, much work has been done to try to characterise the disease however results are conflicting. Most suggest male paddy farmers working in rural areas of the NCP are worst affected, presenting in their fifth decade with end stage renal failure. However, a recent WHO study revealed higher prevalence in females, although more severe renal impairment was more common in men.

Risk factors include inhabiting NCP > five years, inhabiting the 'dry zone', reduced BMI, lower socio-economic class, and exposure to agrochemicals. There has been suggestion of a genetic link although positive family history is limited to one generation, with no evidence of mendelian progression. Epidemiological studies reveal a clustered geographical distribution with areas such as Medawachchiya, Padaviya and Girandurukotte most affected. High prevalence areas encompass a well-developed irrigation system used for agricultural purposes.

Renal biopsies show tubulointerstitial disease with tubular atrophy, interstitial mononuclear cell infiltration, interstitial fibrosis but no immune-complex deposition on immunofluorescence. This supports a toxin-mediated process.

Many aetiologies have been considered including exposure to heavy metals (cadmium, arsenic) and their chelation by herbicides, fluro-aluminium complexes, agricultural pesticides, mycotoxins, and herbal medicines. Selenium deficiency and genetic susceptibility may be predisposing factors. The true aetiology is likely multifactorial.

The multi-system impact of CKDu has yet to be fully realised. Epidemiological and clinical data show that damage to large arteries contributes to the increased cardiovascular risk observed in CKD. Atherosclerosis is the most frequent cause of arterial damage but the medial calcification seen in CKD also leads to arterial stiffening. This stiffening causes elevation in systolic blood pressure, increasing left ventricular workload with the gradual development of LVH, and also a fall in diastolic blood pressure impairing coronary blood flow. Arterial calcification and stiffness are independent predictors of all-cause and cardiovascular mortality in patients with CKD. Arterial stiffness will be compared in CKDu patients, healthy Sri Lankan controls and CKD patients both in Sri Lanka and Scotland.

We will perform a prospective observational study of up to 250 patients with CKDu presenting to renal clinics in Teaching Hospital, Anuradhapura. Patient history, basic anthropometric measurements, and simple non-invasive tests (e.g. blood pressure and arterial stiffness) will be performed. Urine, serum and plasma samples will be collected for quantitative PCR, and further analysis for biomarkers of renal injury, exosomes, proteomics and any DNA-adducts. Patients will be graded using the WHO CKDu grading system. When a renal biopsy is performed, a copy of the light microscopy findings will be obtained. Comparisons of interest will be tested via paired t-tests with statistical significance taken at 5%.

ELIGIBILITY:
CKDu (CKD unknown aetiology) patients:

Inclusion Criteria

* Age 18- 85 years
* Attend CKDu clinic in Anuradhapura or Padavi-Sri Pura
* Evidence of renal dysfunction: proteinuria, raised serum creatinine
* Able to understand information given and happy to give consent

Exclusion Criteria

* Subjects who are on dialysis
* History of diabetes
* History of major cardiac (including MI), respiratory (including asthma & COPD) or neurological disease
* Pregnant
* History of significant hypertension (>140/90mmHg despite anti-hypertensives or >160/100mmHg untreated)
* History of glomerulonephritis or other known cause of renal disease

Inclusion criteria for healthy volunteers:

* Age 18- 85 years
* Present in Anuradhapura teaching hospital as a visitor/carer of patient in ward or at outpatient clinic at either site
* Able to understand information given and happy to give consent

Exclusion criteria for healthy volunteers:

* Age < 18 or >85 years
* Evidence of renal dysfunction: proteinuria, raised serum creatinine
* Evidence of diabetes mellitus, significant hypertension (defined above), glomerulonephritis or other known cause of renal disease.

Inclusion criteria for patients with CKD of known cause:

* Age 18- 85 years
* Attend general renal clinic in Anuradhapura or Padavi-Sri Pura
* Evidence of renal dysfunction: proteinuria, raised serum creatinine
* Known cause renal disease proven by biopsy or strong association such as diabetes mellitus or chronic, severe hypertension.
* Able to understand information given and happy to give consent

Exclusion criteria for patients with CKD of known cause:

* Age < 18 or >85 years
* CKD unknown origin
* Pregnant
* Subjects who are on dialysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending clinics or admitted to hospital during Aug 2014 to Oct 2014 with CKDu (Chronic kidney disease of unknown origin).
  Subjects must be aged 18 to 85 with evidence of renal dysfunction and no other obvious cause noted (see inclusion/exclusion criteria above).
  Control groups will be sought for the measure of arterial stiffness: Sri Lankan CKD of known cause, Sri Lankan healthy volunteers. Our controls will be age, sex and blood pressure matched to the cases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-09; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | 3 months
  Arterial stiffness will be measured using the TensioMed® Arteriograph™. Damage to large arteries contributes to increased cardiovascular risk in CKD. Atherosclerosis is the most frequent cause of arterial damage but medial calcification seen in CKD also leads to arterial stiffening. This stiffening causes elevated systolic blood pressure, increased left ventricular workload and the gradual development of LVH, and also a fall in diastolic blood pressure impairing coronary blood flow. Arterial calcification and stiffness are independent predictors of all-cause and cardiovascular mortality in CKD patients. It is unclear whether the CVD risk associated with CKDu is the same as it is for CKD of known cause. We plan to measure arterial stiffness in both CKD and CKDu patients. We will compare stiffness measurements in CKD of unknown cause with those of a well characterised cohort of CKD patients in Edinburgh. Healthy Sri Lankan volunteers will give an assessment of 'background stiffness'.

SECONDARY OUTCOMES:
Biomarkers of renal disease and DNA adducts | 3 months
  As the aetiology of CKDu remains unknown, we will collect blood and urine samples from a cohort of p to 259 CKDu patients to explore the aetiology further. These samples will be analysed for biomarkers of kidney damage, proteomics, exosomes, and DNA adducts.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eddleston, MA PhD FRCPEdin, Principal Investigator — University of Edinburgh; Neeraj Dhaun, PhD MRCP, Study Director — University of Edinburgh; Sisira Siribaddana, MD FCCP, Study Director — Rajarata University, Sri Lanka
Locations (1):
- Teaching Hospital Anuradhapura, Anuradhapura, North Central Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WHO + Sri Lankan Ministry of Health collaborative study — http://www.biomedcentral.com/1471-2369/14/180
- See also: Oliver JJ, Webb DJ. Noninvasive assessment of arterial stiffness and risk of atherosclerotic events. Arterioscler Thromb Vasc Biol. Apr 1 2003;23(4):554-566 — http://www.ncbi.nlm.nih.gov/pubmed/12615661
- See also: Sarnak MJ, Levey AS et al. Kidney disease as a risk factor for development of cardiovascular disease: a statement from the American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, — http://www.ncbi.nlm.nih.gov/pubmed/14581387